CLINICAL TRIAL: NCT00996775
Title: Implementing Evidence-Based Mental Health Practices in Primary Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIP 62-109
Record Dates: First submitted 2009-10-14; First posted 2009-10-16 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2017-01-02 (Estimated); Status verified 2016-11

CONDITIONS: Alcohol Consumption
Keywords: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking | interventions — Ethanol; Methods; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- standard care only (Active Comparator): standard care only - harmful effects of alcohol use and NIAAA limits
  Interventions: Behavioral: standard care
- Brief alcohol intervention (Experimental): Group receiving brief alcohol intervention
  Interventions: Behavioral: brief alcohol intervention

INTERVENTIONS:
Behavioral: brief alcohol intervention — this intervention consists of brief assessment and feedback
  Arms: Brief alcohol intervention
Behavioral: standard care — education about harmful effects of alcohol use and NIAAA recommended drinking limits
  Arms: standard care only

SUMMARY:
This research study will examine the effectiveness of a brief, computerized motivational intervention plus treatment-as-usual to treatment-as-usual alone for treating alcohol misuse in Veterans presenting to primary care. The investigators aim to recruit 162 Veterans screening positive on the AUDIT-C to participate in this study. Participants will be randomly assigned to one of the two intervention conditions and be asked to complete a baseline assessment and two follow-up assessments conducted at three and six months post treatment. Baseline assessments will be conducted in person by a trained research assistant, while all follow-up interviews will be conducted over the phone. The primary outcome for this clinical trial is the reduction in the number of heavy drinking days. Several secondary outcomes will be collected including health status, depressive symptoms, consequences of drinking, pain symptoms, and distress tolerance. The findings from this study may have large scale implications for how alcohol misuse is treated in primary care. In addition, this study will provide evidence for the feasibility of using the computer as a method for delivering evidence-based mental health interventions in primary care.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age,
* speak and read English,
* U.S. Veteran status,
* screen positive on the AUDIT-C

Exclusion Criteria:

* the presence of any cognitive difficulties that interfere with one's ability to consent to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Cucciare, PhD, Principal Investigator — Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR
Locations (1):
- Central Arkansas Veterans Healthcare System Eugene J. Towbin Healthcare Center, Little Rock, AR, No. Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: Yes
This project will include data from 167 Veterans screening positive for alcohol misuse (without and without posttraumatic stress disorder [PTSD] or depression). Data was collected at three time points including baseline, 3- and 6-month follow-up. The final dataset includes quantitative data including on alcohol consumption, and symptoms of PTSD, and depression. The final dataset will be stripped of identifiers prior to sharing. Release of data for data sharing will occur after publication of the main findings from the dataset. The investigators will make the data and associated documentation available to users under our own auspices by mailing an encrypted hard-drive to users. A data-sharing agreement must be signed that accounts for (1) commitment to using the data only for research; (2) IRB approval at the host institution, (3) a plan for securing the data using appropriate technology, and (4) an agreed upon plan to destroy or return the data upon completion.

REFERENCES:
- [Result] Cucciare MA, Ghaus S. A Web-based intervention for alcohol misuse in VA primary care. Psychiatr Serv. 2012 Mar;63(3):292. doi: 10.1176/appi.ps.20120p292. No abstract available. PMID 22388536
- [Result] Cucciare MA, Boden MT, Weingardt KR. Brief alcohol counseling improves mental health functioning in veterans with alcohol misuse: results from a randomized trial. J Affect Disord. 2013 May;147(1-3):312-7. doi: 10.1016/j.jad.2012.11.028. Epub 2012 Dec 6. PMID 23218847
- [Result] Cucciare MA, Weingardt KR, Ghaus S, Boden MT, Frayne SM. A randomized controlled trial of a web-delivered brief alcohol intervention in Veterans Affairs primary care. J Stud Alcohol Drugs. 2013 May;74(3):428-36. doi: 10.15288/jsad.2013.74.428. PMID 23490572

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Group receiving treatment-as-usual.
  Treatment-as-Usual: Treatment-as-usual for positive AUDIT-C screens conducted in the GMC at the VA Palo Alto Health Care System.
- Arm 2: Group receiving treatment-as-usual plus a brief alcohol intervention
  brief alcohol intervention: computer-delivered intervention consisting of an assessment and individualized feedback component.
  Treatment-as-Usual: Treatment-as-usual for positive AUDIT-C screens conducted in the GMC at the VA Palo Alto Health Care System.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 78 | 89
Completed | 67 | 75
Not Completed | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 78 | 89 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (15.9) | 60.8 (14.1) | 59.0 (15.0)
Gender [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 68 | 79 | 147

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Percentage of Heavy Drinking Days
Description: reduction in the percentage of heavy drinking days over the prior 30-days.
  a heavy drinking day was defined as drinking above gender-matched NIAAA drinking limits (e.g., greater than 4 drinks on one occasion for men).
Time Frame: baseline to six-month follow-up
Measure: Mean (Standard Deviation); unit: percentage of heavy drinking days
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 78 | 89
percentage of heavy drinking days | 14.0 (25.0) | 11.0 (23.0)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes